CLINICAL TRIAL: NCT04746495
Title: Effect of Eplerenone on Novel Biomarkers of Mineralocorticoid Receptor Activation (ENOVA)
Acronym: ENOVA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Issues relate to COVID-19 and staffing challenges, as well as very tight finances.
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, J Brian Byrd, MD, MS, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HUM00170418; 1K23HL128909-01A1 (NIH)
Record Dates: First submitted 2021-01-12; First posted 2021-02-09 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hypertension
Keywords: mineralocorticoid; mineralocorticoid receptor; aldosterone; eplerenone; blood pressure
MeSH Terms: conditions — Hypertension | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: * Lab results will be reviewed by an un-blinded co-investigator.
  * Dose adjustments will be done by an un-blinded co-investigator who is licensed to prescribe the study drug.
  * The study blind will be broken on completion of the clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will be randomized to receive 4 weeks of placebo and then 4 weeks of Eplerenone.
  Interventions: Drug: Placebo
- Eplerenone (Experimental): Participants will be randomized to receive 4 weeks of Eplerenone and then 4 weeks of Placebo.
  Interventions: Drug: Eplerenone 50mg

INTERVENTIONS:
Drug: Placebo — Participants will go through a 2-week wash-in period. During the wash-in period, the participant will be asked not to take their usual antihypertensive medications for their mild hypertension. After the 2-week wash-in period, the participants will begin a 4-week treatment period and will take a placebo once a day for 4 weeks. After the 4 weeks, the participants will have a 2-week wash-out period where they will be off the study treatment. After the 2-week wash-out period, the participants will begin the Eplerenone treatment for another 4 weeks.
  Arms: Placebo
Drug: Eplerenone 50mg — Participants will go through a 2-week wash-in period. During the wash-in period, the participant will be asked not to take their usual antihypertensive medications for their mild hypertension. After the 2-week wash-in period, the participants will begin a 4-week treatment period of Eplerenone for 4 weeks. After the 4 weeks, the participants will have a 2-week wash-out period where they will be off the study treatment. After the 2-week wash-out period, the participants will then begin the Placebo treatment for another 4 weeks.
  Arms: Eplerenone

SUMMARY:
This blinded cross-over clinical trial will enroll participants with mild stage 1 hypertension to evaluate whether urinary extracellular transcript abundance predicts response to an mineralocorticoid receptor (MR) antagonist, eplerenone.

Eligible participants will have a 2 week wash-in period followed by 4 weeks of treatment with placebo or eplerenone. There will be a 2 week wash out period from study medications and then participants will take the other drug (placebo or eplerenone) for 4 weeks. In addition, participants will also provide urine and blood samples during the trial, have physical assessments, and be monitored for safety.

ELIGIBILITY:
Inclusion Criteria:

* History of mild stage 1 systemic hypertension as defined by:

  1. Systolic blood pressure (SBP) ≥ 140 millimeters of Mercury (mmHg) or diastolic blood pressure (DBP) ≥ 90 mmHg on 2 occasions and
  2. Treatment with 1-2 antihypertensive medications (stable dose for 6 weeks)

     Exclusion Criteria:
* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Stage 2 hypertension (history of blood pressure ≥ 160/100 mmHg)
* History of hypertensive urgency, hypertensive crisis, or hospitalizations for hypertension
* Current mineralocorticoid antagonist use
* Type II Diabetes with microalbuminuria
* Primary adrenal insufficiency
* Current glucocorticoid use
* Electrolyte abnormality on baseline laboratory assessment
* Current potassium supplementation
* Positive test for leukocyte esterase on urinalysis
* Creatinine clearance < 50 mL/min on baseline laboratory assessment
* Hyperkalemia
* Potassium-sparing diuretics (e.g., amiloride, spironolactone, or triamterene)
* Serum potassium >5.0 milliequivalents per liter (mEq/L) on baseline laboratory assessment
* Current use of strong CYP3A4 inhibitors (some include: ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir, and nelfinavir).
* Serum creatinine > 1.5 mg/dL in males on baseline laboratory assessment
* Serum creatinine > 1.3 mg/dL in females
* Current beta blocker use
* Any other condition thought by the Principal Investigator to place the participant at increased risk of injury during the clinical trial or compromise the scientific integrity of the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Reverse transcriptase quantitative polymerase chain reaction (RT-qPCR) Cycle threshold (Ct) value of mineralocorticoid receptor-regulated gene messenger ribonucleic acid (mRNA) | Week 6 (after first study treatment)
  Cycle threshold of urinary mRNA biomarker following treatment with placebo and following treatment with eplerenone will be measured using RT-qPCR.
RT-qPCR Ct value of mineralocorticoid receptor-regulated gene mRNA | Week 12 (after second study treatment)
  Cycle threshold of urinary mRNA biomarker following treatment with placebo and following treatment with eplerenone will be measured using RT-qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: J Brian Byrd, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
We will de-identify participant information and will share it with a trusted repository, such as National Institutes of Health (NIH) Figshare or The Inter-university Consortium for Political and Social Research (ICPSR).
  We will de-identify and share data obtained from analyzing urinary mRNA biomarkers and measuring the systolic and diastolic blood pressure following consumption of a high-sodium and low-sodium diet. Additionally, specific lab values that support the validity and quality of the study treatment will be shared in a trusted repository.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified data will be deposited into a repository within 1 year of the conclusion of the study.
Access Criteria: No additional access restrictions will be placed on the de-identified data, beyond those required by the repository to access or download the data.